CLINICAL TRIAL: NCT02845063
Title: Effects of ACE Genotype on Muscular and Functional Adaptations Following a Cardiovascular Rehabilitation Program
Brief Title: Effect of ACE Genotype on Cardiovascular Rehabilitation
Acronym: ACE-REHAB
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated
Sponsor: Balgrist University Hospital (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: W 549 ACE-REHAB; KEK-ZH-Nr. 2014-0319 (Other: Ethics Committee of the Canton Zurich, Switzerland)
Record Dates: First submitted 2015-11-27; First posted 2016-07-27 (Estimated); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Disease
Keywords: muscle plasticity; exercise; rehabilitation; perfusion; ACE; genotype; hypertension; molecular biology
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- concentric cardiovascular rehabilitation (Experimental): Heart patients under ACE inhibitor intake will be enrolled in the intervention 'concentric cardiovascular training' and evaluated by the intervention 'ACE genotyping'
  Interventions: Behavioral: concentric cardiovascular training; Genetic: ACE genotyping
- eccentric cardiovascular rehabilitation (Experimental): Heart patients under ACE inhibitor intake will be enrolled in the intervention 'eccentric cardiovascular training' and evaluated by the intervention 'ACE genotyping'
  Interventions: Behavioral: eccentric cardiovascular training; Genetic: ACE genotyping
- concentric cardiovascular training (Active Comparator): Healthy subjects will be enrolled in the intervention 'concentric cardiovascular training' and evaluated by the intervention 'ACE genotyping'
  Interventions: Behavioral: concentric cardiovascular training; Genetic: ACE genotyping
- eccentric cardiovascular training (Active Comparator): Healthy subjects will be enrolled in the intervention 'eccentric cardiovascular training' and evaluated by the intervention 'ACE genotyping'
  Interventions: Behavioral: eccentric cardiovascular training; Genetic: ACE genotyping

INTERVENTIONS:
Behavioral: concentric cardiovascular training — Subjects will carry out 8 weeks of cardiovascular training by an interval type of protocol that includes a high repetition number of concentric type contractions on a softrobotic device.
  Arms: concentric cardiovascular rehabilitation; concentric cardiovascular training
Behavioral: eccentric cardiovascular training — Subjects will carry out 8 weeks of cardiovascular training by an interval type of protocol that includes a high repetition number of eccentric type contractions on a softrobotic device.
  Arms: eccentric cardiovascular rehabilitation; eccentric cardiovascular training
Genetic: ACE genotyping — Subjects will be genotyped for the ACE-I/D gene polymorphism.

SUMMARY:
The study aims to systematically investigate the interaction between training modality, ACE genotype and disease in heart patients whom complete a cardiovascular rehabilitation program. This is carried out with the goal to improve the benefit of cardiovascular rehabilitation for the patient by maximising adjustments in muscle structure and function with the intervention. A population of healthy individuals will be recruited who will carry out the same training program, in order to compare the training effects respective to the general population.

DETAILED DESCRIPTION:
Pharmacological inhibition of angiotensin converting enzyme modifies exercise-induced pro-angiogenic and mitochondrial gene transcript expression. Exercise-induced muscle plasticity importantly interacts with the insertion/deletion genotype of ACE and the training modality and intensity. The aim of this study is to systematically investigate the interaction between training modality, ACE genotype and disease in heart patients whom complete a cardiovascular rehabilitation program.

There are two training modalities being used: The first modality involves cardiovascular training by an interval type of protocol that includes a high repetition number of shortening (i.e. concentric) type contractions on a softrobotic device. The second modality includes a high repetition number of lengthening (i.e. eccentric) type contractions on a softrobotic device. In both training modalities the same muscle groups are exercised over the same range of motion, with the same speed of movement, but with widely differing pedal force. Total absolute external mechanical work will be matched.

In order to assess the baseline values and the effect size of the muscle and training adjustments made, healthy male and female volunteers will be included who are matched with respect to age and sex to the patient population and undergo the same training program.

ELIGIBILITY:
Patient group inclusion criteria:

* stable coronary heart patients/heart patients without ischemia
* Left ventricular ejection fraction > 50%
* Drug therapy with ACE inhibitors
* V̇O2peak <86% of the medical reference value Voluntary participation
* Written informed consent of the subject to participate in the study

exclusion criteria:

* relevant valvular heart disease
* arterial hypertension (blood pressure at rest> 140/90)
* arrhythmogenic cardiomyopathy
* ACE inhibitor intolerance
* contraindication for ethical reasons
* known or suspected non-compliance with the curriculum
* smoker
* drug or alcohol disease
* inability of the patient to follow the study procedures (e.g. because of language problems, mental illness, dementia)
* participation in another clinical trial within the last 30 days prior to confinement and during the study
* other, clinically significant comorbidities (cardiac arrhythmia, renal insufficiency, hepatic dysfunction, connective tissue disease [Marfan syndrome, Ehlers-Danlos syndrome])

Healthy subject group inclusion criteria:

* inconspicuous ECG under exercise (persons in whom the exercise ECG is abnormal will be referred for a cardiological evaluation recessed to the University Hospital Zurich)
* V̇O2peak <50 ml O2 min-1 kg-1
* Voluntary participation
* Written informed consent of the subject to participate in the study

exclusion criteria:

* relevant valvular heart disease
* arterial hypertension (blood pressure at rest> 140/90)
* arrhythmogenic cardiomyopathy
* ACE inhibitor intolerance
* contraindication for ethical reasons
* known or suspected non-compliance with the curriculum
* smoker
* drug or alcohol disease
* inability of the patient to follow the study procedures (e.g. because of language problems, mental illness, dementia)
* participation in another clinical trial within the last 30 days prior to confinement and during the study
* other, clinically significant comorbidities (cardiac arrhythmia, renal insufficiency, hepatic dysfunction, connective tissue disease [Marfan syndrome, Ehlers-Danlos syndrome])

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
ACE I/D genotype | 975 days: May 2016-January 2019
  Genotype of the assessed insertion/deletion gene polymorphism of angiotensin converting enzyme ACE, i.e. ACE-II, ACE-ID or ACE-DD.
Molecular muscle characteristics - mRNA | 975 days: May 2016-January 2019
  • mRNA expression of VEGF, HIF-1a, HIF-1b, tenascin-C, Angpt1, Angpt1R, neuropilin, midkine, restin, COX4-1, COX4I-2, CPTI, LPL, LIPE, FATP, CD36 [relative expression per 28S rRNA]
Molecular muscle characteristics- protein | 975 days: May 2016-January 2019
  • Protein content of FAK, FRNK, p70S6K, mTOR, JNK, NDUFA9, SDH, UQCRC1, COX4I1, COX4I2, ATP5A1, VEGF, HIF-1a, CD31, MHC-1, MHC-2A, MHC-2X, MyoD, myogenin, CaMKII [pixel counts per actin]
Molecular muscle characteristics- phosphorylation | 975 days: May 2016-January 2019
  • Phosphorylation of proteins phospho-Y397- FAK, phospho-T421/S424-P70S6K, phospho -T183/Y185-JNK, phospho-S2448-mTOR [pixel counts per actin]
Molecular muscle characteristics- ACE | 975 days: May 2016-January 2019
  • ACE activity [fmol min-1]
Cellular muscle characteristics - fiber type % | 975 days: May 2016-January 2019
  • Distribution of type I, IIA and IIX fibers [%]
Cellular muscle characteristics - fiber area % | 975 days: May 2016-January 2019
  • Area percentage of type I, IIA and IIX fibers [% area]
Cellular muscle characteristics - fiber type CSA | 975 days: May 2016-January 2019
  • Cross sectional area of type I, IIA and IIX fibers [micrometer2]
Cellular muscle characteristics - Capillary density | 975 days: May 2016-January 2019
  • Capillary density [capillaries micrometer-2]
Cellular muscle characteristics - Capillary-to-fiber ratio | 975 days: May 2016-January 2019
  • Capillary-to-fiber ratio
Functional muscle characteristics - Maximal Power | 975 days: May 2016-January 2019
  • Maximal power during ramp test on ergometer [Watt]
Functional muscle characteristics - Critical Power | 975 days: May 2016-January 2019
  • Critical power in ramp test on ergometer [Watt]
Functional muscle characteristics - Real Power | 975 days: May 2016-January 2019
  • Real Power as estimated on the soft robotic device [Watt]
Functional muscle characteristics - Reactive Power | 975 days: May 2016-January 2019
  • Reactive Power as estimated on the soft robotic device [Watt]
Functional muscle characteristics - Negative Power | 975 days: May 2016-January 2019
  • Negative Power as estimated on the soft robotic device [Watt]
Functional muscle characteristics - Maximal force | 975 days: May 2016-January 2019
  • Maximal force during the reactive power test on the soft robotic device [Newton]
Functional muscle characteristics - Maximal velocity | 975 days: May 2016-January 2019
  • Maximal velocity during the reactive power test on the soft robotic device [m sec-1]
Functional muscle characteristics - Rate of force development | 975 days: May 2016-January 2019
  • Rate of force development as estimated during the Real Power test on the soft robotic device [meter sec-2]
Muscle metabolism - muscle oxygenation ramp | 975 days: May 2016-January 2019
  • Muscle oxygenation (m. vastus lateralis, m. gastrocnemius, m. gluteus maximus) during ramp test on ergometer [%]
Muscle metabolism - muscle oxygenation robot exercise | 975 days: May 2016-January 2019
  • Muscle oxygenation (m. vastus lateralis, m. gastrocnemius, m. gluteus maximus) during exercise on soft robot [%]
Muscle metabolism - hemoglobin ramp | 975 days: May 2016-January 2019
  • Total hemoglobin during ramp test on ergometer [%]
Muscle metabolism - hemoglobin robot exercise | 975 days: May 2016-January 2019
  • Total hemoglobin during exercise on soft robot [%]
Muscle metabolism - lipid compounds | 975 days: May 2016-January 2019
  • Concentration of lipid compounds in m. vastus lateralis muscle during exercise on soft roboter
Muscle metabolism - metabolites | 975 days: May 2016-January 2019
  • Concentration of metabolites in m. vastus lateralis muscle during exercise on soft roboter
Muscle metabolism - serum glucose | 975 days: May 2016-January 2019
  • Concentration of glucose in serum during ramp test on ergometer [mmol l-1]
Muscle metabolism - serum lactate | 975 days: May 2016-January 2019
  • Concentration of lactate in serum during ramp test on ergometer [mmol l-1]
Cardiovascular function - Heart rate rest | 975 days: May 2016-January 2019
  • Heart rate at rest [beats per minute]
Cardiovascular function - Heart rate ramp | 975 days: May 2016-January 2019
  • Heart rate in ramp test on ergometer [beats per minute]
Cardiovascular function - cardiac output | 975 days: May 2016-January 2019
  • Cardiac output [L min-1]
Cardiovascular function - ejection fraction | 975 days: May 2016-January 2019
  • Ejection fraction
Cardiovascular function - Maximal oxygen uptake | 975 days: May 2016-January 2019
  • Maximal oxygen uptake (VO2max) during ramp test on ergometer [ml O2 min-1 kg-1]
Cardiovascular function - ventilation | 975 days: May 2016-January 2019
  • Ventilation during ramp test on ergometer [L min-1]
Cardiovascular function - ventilation frequency | 975 days: May 2016-January 2019
  • Ventilation frequency ramp test on ergometer [min-1]
Cardiovascular function - respiration quotient | 975 days: May 2016-January 2019
  • Respiration quotient during ramp test on ergometer [ L O2 inspired / L CO2 expired]
Cardiovascular function - endurance | 975 days: May 2016-January 2019
  Time-to-exhaustion in constant load on ergometer [seconds]

CONTACTS AND LOCATIONS:
Overall Officials: Walter O Frey, MD, Principal Investigator — Balgrist University Hospital, Move>med, Swiss Olympic Center, Zurich, Switzerland; Christian M Schmied, MD, Principal Investigator — Cardiology, University Hospital Zurich, Zurich, Switzerland
Locations (2):
- Switzerland (2):
  - Balgrist University Hospital, Zurich
  - University Hospital Zurich, Zurich

REFERENCES:
- [Background] van Ginkel S, Ruoss S, Valdivieso P, Degens H, Waldron S, de Haan A, Fluck M. ACE inhibition modifies exercise-induced pro-angiogenic and mitochondrial gene transcript expression. Scand J Med Sci Sports. 2016 Oct;26(10):1180-7. doi: 10.1111/sms.12572. Epub 2015 Sep 26. PMID 26407530
- [Background] van Ginkel S, Amami M, Dela F, Niederseer D, Narici MV, Niebauer J, Scheiber P, Muller E, Fluck M. Adjustments of muscle capillarity but not mitochondrial protein with skiing in the elderly. Scand J Med Sci Sports. 2015 Aug;25(4):e360-7. doi: 10.1111/sms.12324. Epub 2014 Sep 28. PMID 25262765
- [Background] Mathes S, van Ginkel SL, Vaughan D, Valdivieso P, Flück M, Gene-pharmacologial effects on exercise-induced muscle gene expression in healthy men. Anat Physiol 2015, S5.
- [Background] van Ginkel S, de Haan A, Woerdeman J, Vanhees L, Serne E, de Koning J, Fluck M. Exercise intensity modulates capillary perfusion in correspondence with ACE I/D modulated serum angiotensin II levels. Appl Transl Genom. 2015 Mar 27;4:33-7. doi: 10.1016/j.atg.2015.03.002. eCollection 2015 Mar. PMID 26937347
- [Background] Vaughan D, Huber-Abel FA, Graber F, Hoppeler H, Fluck M. The angiotensin converting enzyme insertion/deletion polymorphism alters the response of muscle energy supply lines to exercise. Eur J Appl Physiol. 2013 Jul;113(7):1719-29. doi: 10.1007/s00421-012-2583-6. Epub 2013 Feb 9. PMID 23397151
- [Derived] Fitze DP, Franchi M, Popp WL, Ruoss S, Catuogno S, Camenisch K, Lehmann D, Schmied CM, Niederseer D, Frey WO, Fluck M. Concentric and Eccentric Pedaling-Type Interval Exercise on a Soft Robot for Stable Coronary Artery Disease Patients: Toward a Personalized Protocol. JMIR Res Protoc. 2019 Mar 27;8(3):e10970. doi: 10.2196/10970. PMID 30916659
- See also: van Ginkel et al, 2015 — http://dx.doi.org/10.1016/j.atg.2015.03.002